CLINICAL TRIAL: NCT05528484
Title: Effect of ERAS Nursing on Self-reported Outcomes of Patients Undergoing Minimally Invasive Lung Cancer Surgery
Brief Title: Self-reported Outcomes of Patients in ERAS Nursing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ERAS (PRO)-based study
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-08

CONDITIONS: Enhanced Recovery After Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Experimental): the patients accepting eras nursing protocol ;
  Interventions: Procedure: ERAS nursing
- non-eras group (Active Comparator): the patients not accepting eras nursing protocol ;
  Interventions: Procedure: non eras nursing

INTERVENTIONS:
Procedure: ERAS nursing — Patients were given education before surgery, fluid and anesthetic drug management during surgery, early ambulation, fluid management and early feeding after surgery, etc
  Arms: ERAS group
Procedure: non eras nursing — Patients were under the routine management without eras protocol
  Arms: non-eras group

SUMMARY:
We aimed to evaluate the effect of ERAS nursing program on self-reported outcomes of patients undergoing minimally invasive lung cancer surgery, and compared the differences in length of hospital stay, complications, and readmission rate between ERAS and non-ERAS nursing programs

ELIGIBILITY:
Inclusion Criteria:

* ≥18years,Minimally invasive elective surgery,cooperate

Exclusion Criteria:

* Pneumonectomy was performed and converted to open surgery

Surgery intensive care, unable to cooperate (language

Speech disorders, psychopathology)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported Outcomes of Patients(PRO) | at baseline, daily after surgery, and weekly up to 4 after discharge weekly.
  Use MD Anderson Symptom Checklist - Lung Cancer Symptom to measure severity and functional status

SECONDARY OUTCOMES:
length of stay (LOS), postoperative cardiopulmonary complications (CPC) and readmission rate (READM) | From admission to one month after the patient's discharge
  length of stay (LOS), postoperative cardiopulmonary complications (CPC) and readmission rate (READM)

CONTACTS AND LOCATIONS:
Locations (1):
- The second hospital of shandong university, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided